CLINICAL TRIAL: NCT00366704
Title: A Multicenter, Randomized, Double-blind, Parallel-group Fixed-dose Study of the Effect on Weight of Bifeprunox Versus Risperidone in the Treatment of Outpatients With Schizophrenia.
Brief Title: Study Comparing Bifeprunox to Risperidone in Treatment of Outpatients With Schizophrenia With Weight as Primary Endpoint
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Collaborators: Solvay Pharmaceuticals (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3168A1-313; B3101009 (Other: Pfizer)
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2008-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — bifeprunox; Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: bifeprunox
- B (Active Comparator)
  Interventions: Drug: risperidone

INTERVENTIONS:
Drug: bifeprunox — .25mg titrate up to 20mg/day (week 1) then 30mg/day (weeks 2-8)
  Arms: A
Drug: risperidone — 4mg, QD, 8 week treatment
  Arms: B

SUMMARY:
The purpose of this study is to determine the effect of bifeprunox or risperidone on the body weight of patients with schizophrenia.

ELIGIBILITY:
Inclusion criteria:

* Current treatment of at least 3 months with risperidone.
* Primary diagnosis of schizophrenia.
* Total Positive and Negative Symptoms Scale (PANSS) score < or = 70 at screening and baseline.

Exclusion criteria:

* Psychiatric diagnosis other than schizophrenia as assessed by the modified Mini International Neuropsychiatric Interview (MINI) and considered by the investigator to be the primary psychiatric diagnosis.
* History or presence of clinically significant cardiovascular, endocrine, hepatic, renal or other medical disease that might be detrimental to the subject or confound the study.
* History of any suicide attempt within 3 years of day 1 or significant immediate risk of violence or suicidality.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2006-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
The primary analysis will be the change from baseline on body weight at the final evaluation. | 8 weeks

SECONDARY OUTCOMES:
Secondary outcomes include: Change from baseline in triglyceride level, Change from baseline in waist circumference, and Change from baseline in total Positive and Negative Syndrome Scale (PANSS) score. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (55):
- United States (55):
  - Little Rock, Arkansas
  - Anaheim, California
  - Boynton Beach, California
  - Costa Mesa, California
  - Escondido, California
  - Garden Grove, California
  - Glendale, California
  - Huntington Beach, California
  - La Mesa, California
  - National City, California
  - Oceanside, California
  - Paramount, California
  - Rosemead, California
  - San Diego, California
  - Santa Ana, California
  - New London, Connecticut
  - Fort Lauderdale, Florida
  - Jacksonville, Florida
  - North Miami, Florida
  - St. Petersburg, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Marietta, Georgia
  - Coevr d'Alene, Idaho
  - Chicago, Illinois
  - Hoffman Estates, Illinois
  - Joliet, Illinois
  - Naperville, Illinois
  - Lake Charles, Louisiana
  - Gaithersburg, Maryland
  - Pittsfield, Massachusetts
  - Worcester, Massachusetts
  - Flowood, Mississippi
  - St Louis, Missouri
  - North Platte, Nebraska
  - Cherry Hill, New Jersey
  - Clementon, New Jersey
  - Rochester, New York
  - Staten Island, New York
  - Butner, North Carolina
  - Morehead City, North Carolina
  - Beachwood, Ohio
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - East Stroudsberg, Pennsylvania
  - Jenkintown, Pennsylvania
  - Norristown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Cordova, Tennessee
  - Memphis, Tennessee
  - Austin, Texas
  - DeSoto, Texas
  - Irving, Texas
  - San Antonio, Texas